CLINICAL TRIAL: NCT06691698
Title: Evaluation of The Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach for Adolescents With Mild Intellectual Disability
Brief Title: Evaluation of CO-OP for Adolescents With Mild Intellectual Disability
Acronym: CO-OPIF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Landstinget i Värmland (Other); Göteborg University (Other); Stiftelsen Sunnerdahls Handikappfond (Other); Stiftelsen Sävstaholm (Unknown); Majblommans riksförbund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORU 2024-02873-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Intellectual Disability, Mild
Keywords: adolescents; executive function; metacognition; mild intellectual disability; occupational therapy; occupational performance; person-centered intervention; self-efficacy
MeSH Terms: conditions — Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Masking Description: One of the outcomes will be assessed using video from baseline, post and 6 months post intervention, and the assessor of those videos will be blinded to the order and have no knowledge about the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO-OP for adolescents with mild intellectual disability (Experimental): CO-OP intervention during 10 weeks. Outcomes measures at baseline, directly after and 6 months after intervention
  Interventions: Other: The Cognitive Orientation to Daily Occupational Performance Approach

INTERVENTIONS:
Other: The Cognitive Orientation to Daily Occupational Performance Approach — CO-OP is a client-centred, performance-based, problem-solving focused, occupation-focused and occupation-based intervention. In CO-OP the person is guided to use a meta-cognitive strategy to find his or her own strategies for specific activities. The main purpose is to enable meta-cognitive thinking in every day activities, leading to enhanced self-efficacy, occupational performance and independency.
  Other Names: CO-OP

SUMMARY:
Intellectual disability (ID) affects a person throughout life and includes difficulties to manage what is expected in everyday life based on age. One difficulty is to create strategies for and solve problems related to everyday occupations. Treatment options with good evidence to enhance occupational performance for persons with ID are limited. The Cognitive Orientation to Daily Occupational Performance (CO-OP) is an approach with good evidence within other diagnostic groups, i.e. adolescents with cerebral palsy. CO-OP has a unique person-centered approach where the person chooses his/her own goals and creates his/her own strategies to reach them. Initial research shows potential for CO-OP with adolescents with ID, although due to scientific flaws there is still a lack of evidence regarding feasibility and effectiveness for adolescents with ID. Based on the results with other diagnostic groups and clinical knowledge and experience, CO-OP can be assumed to be feasible and effective for adolescents with ID and to have a long term effect transferred to everyday life in a way other treatment options do not.

The aim of the project is to describe and evaluate CO-OP for adolescents with mild ID. Participants will be adolescents aged 13-17 and their parents. The project is designed as a feasibility study with two qualitative, one quantitative and one mixed method data collection. The quantitative data will be ordinal and nominal data from observational and self-assessment assessments. The mixed methods include comparison between filmed sessions and the CO-OP manual, use of field notes to analyse fidelity and needs for adaptations, and comparison between the CO-OP manual and policy documents. The qualitative outcome will be experiences by the adolescents and perceptions of CO-OP by parents.

ELIGIBILITY:
Study I-II

Inclusion criteria

* 13-17 years
* Diagnosed mild intellectual disability
* Motivation to reach self-selected goals
* Ability to identify those goals
* Possibility to meet once a week for ten weeks
* Access to a parent or significant other for support during intervention

Exclusion criteria:

* Movement related diagnosis (i.e. cerebral palsy or neuro muscular diseases)
* Diagnosed attention deficit hyperactivity disorder/attention deficit disorder (ADHD/ADD) or autism spectrum disorder
* Progressive diagnoses
* Need for language interpreting
* Need for alternative and augmentative communication (i.e. pictures or signs).

Study III

Inclusion criteria:

* 13-17 years
* Diagnosed mild intellectual disability
* Completed CO-OP intervention or at lest half way trough the intervention
* Opportunity to meet physically for an interview with in a month post and 6 months post intervention.
* CO-OP intervention done with high fidelity to CO-OP format with a CO-OP therapist that has written field notes, preferrably recruited from study I-II.

Exclusion criteria:

* Movement related diagnosis (i.e. cerebral palsy or neuro muscular diseases)
* Diagnosed attention deficit hyperactivity disorder/attention deficit disorder (ADHD/ADD) or autism spectrum disorder
* Progressive diagnoses
* Need for language interpreting
* Need for alternative and augmentative communication (i.e. pictures or signs).

Study IV

Inclusion criteria:

* Parents with legal guardianship that lives full- or part time with an adolescent reaching the inclusion criteria for study I who has completed CO-OP within or out of the project
* Opportunity to meet physically for an interview with in a month post and 6 months post the adolescent's completed, or at least half way through, CO-OP intervention.

Exclusion criteria:

* Need for language interpreting
* Need for alternative and augmentative communication (i.e. pictures or signs)
* Irregular and brief living with the adolescent comparable to less than half-time and therefore does not observe the adolescent's occupational performance enough to answer the interview questions.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure - performance | Baseline, up to 4 weeks post intervention and 6 months post intervention
  Self-rated occupational performance in four chosen goal activities, rated 1-10
Change in Canadian Occupational Performance Measure - satisfaction | Baseline, up to 4 weeks post intervention and 6 months post intervention
  Self-rated satisfaction with performance in four chosen goal activities, rated 1-10
Change in Performance Quality Rating Scale - occupational performance quality | Baseline, up to 4 weeks post intervention and 6 months post intervention
  Observed performance quality during performing four chosen goal activities thas is filmed and rated 1-10.

SECONDARY OUTCOMES:
Change in General Self-Efficacy Scale - self-efficacy | Baseline, up to 4 weeks post intervention and 6 months post intervention
  Self-rated self-efficacy, 10 statements rated 1-4.
Experiences of CO-OP as a patient - qualitative | Up to 4 weeks post intervention and 6 months post intervention
  Qualitative semi-structured interviews analyzed using qualitative content analysis.
Perceptions of CO-OP as a parent of a patient - qualitative | Up to 4 weeks post intervention and 6 months post intervention
  Qualitative semi-structured interviews analyzed using phenomenographic analysis

OTHER OUTCOMES:
Feasibility: Acceptability | Up to 4 weeks post intervention and 6 months post intervention
  Acceptability will be evaluated by structured interviews. The interview consists of five yes/no questions and a 10 point scale on how much effort the CO-OP intervention required. Data will be on nominal and ordinal level.
Feasibility: Possible expansion to a new group | 2024-2025
  Qualitative text analysis in which contents of the CO-OP manual will be compared with norms and values in the national policy documents for children and youth habilitation. This is carried out to evaluate whether it would be possible to expand this intervention to a new group of patients (adolescents with mild intellectual disability). The data collection is not related to the individual participants.
Feasibility: Adaptation | Up to 1 year after intervention.
  Whether the CO-OP approach needs any adaptations in order to be feasible for adolescents with mild intellectual disability will be evaluated. This will be done by collecting field notes written by CO-OP therapists and a text analysis with descriptive comparison between notes and the CO-OP manual.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Holmefur, PhD, Principal Investigator — Örebro University, Sweden
Locations (2):
- Sweden (2):
  - Region Skåne, Kristianstad, Skåne County
  - Region Värmland, Karlstad, Värmland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project presentation at Orebro University website. — https://www.oru.se/forskning/forskningsprojekt/fp/?rdb=p2711